CLINICAL TRIAL: NCT00656084
Title: A Phase II Study of Gemzar, Novantrone and Rituxan in Relapsed or Refractory Mantle Cell Lymphoma (MCL) (B9E-US-X436)
Brief Title: Ph2 Gem/Nov/Rituxan Rel/Ref MantleCell
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Dr. Lawrence Garbo, Principal Investigator, US Oncology Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-026
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Results first posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-09

CONDITIONS: Relapsed or Refractory Mantle Cell Lymphoma (MCL)
MeSH Terms: conditions — Recurrence; Lymphoma, Mantle-Cell | interventions — Gemcitabine; Mitoxantrone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental arm (Experimental): Patients will be treated a maximum of 8 cycles or until the patient has evidence of a response, progressive disease, or until intolerable toxicity develops. Patients with a complete response will receive an additional 2 cycles of treatment (not to exceed 8 cycles). Drug order is gemcitabine, mitoxantrone, and rituximab.
  Interventions: Drug: gemcitabine; Drug: mitoxantrone; Drug: rituximab

INTERVENTIONS:
Drug: gemcitabine — 900 mg/m2 on Days 1 and 8 of each 21-day cycle The order of administration will be: Gemzar-->Novantrone-->Rituxan.
  Other Names: Gemzar
Drug: mitoxantrone — Novantrone 10 mg/m2on Day 1. The order of administration will be:
  Gemzar-->Novantrone-->Rituxan.
  Other Names: Novantrone
Drug: rituximab — Rituxan 375 mg/m2 on Day 1. The order of administration will be:
  Gemzar-->Novantrone-->Rituxan.
  Other Names: Rituxan

SUMMARY:
To determine the efficacy (response rate) produced by the combination of Gemzar, Novantrone, and Rituxan in relapsed or refractory MCL

ELIGIBILITY:
Inclusion Criteria:

* Stage III or IV, histologically confirmed relapsed or refractory MCL as reviewed by the SI
* Is CD20 positive (by immunohistochemistry or FACS)
* Is Cyclin D positive (by immunohistochemistry or FACS)
* Has received prior chemotherapy (required minimum of 1 prior therapies)
* Has received prior treatment with Rituxan
* Has an ECOG Performance Status (PS) 0-2
* Is greater than or equal to 18 years of age
* Has appropriate laboratory values (please refer to protocol for specific laboratory values)
* If a history of cardiac disease is indicated, patient has an LVEF greater than or equal to 50% (MUGA)
* Has a negative serum pregnancy test within 7 days prior to registration (female patients of childbearing potential)
* If fertile, patient (male or female) has agreed to use an acceptable method of birth control to avoid pregnancy for the duration of the study and for a period of 2 months thereafter
* Has signed a Patient Informed Consent Form
* Has signed a Patient Authorization Form

Exclusion Criteria:

* Has other lymphomas not classified as MCL
* Has had prior treatment with Gemzar and/or Novantrone
* A history of known hypersensitivity to Gemzar, Novantrone, Rituxan, or any component of these drugs
* Has a history of hypersensitivity to murine-cell derived therapeutics
* Has a LVEF indicative of a cardiac condition (LVEF < 50%)
* Is receiving concurrent immunotherapy
* Has evidence of CNS involvement
* Has a serious uncontrolled intercurrent medical or psychiatric illness, including serious infection
* Has a history of other malignancy within the last 5 years (except cured basal cell carcinoma of skin and carcinoma insitu of uterine cervix), which could affect the diagnosis or assessment of any of the study drugs
* Is a pregnant or nursing woman
* Is unable to comply with requirements of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-12; Primary Completion 2007-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Garbo, MD, Principal Investigator — US Oncology Research

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemzar + Novantrone + Rituxan: Gemzar, Novantrone, and Rituxan in relapsed or refractory mantle cell lymphoma (MCL)
Period: Overall Study
Arm/Group | Gemzar + Novantrone + Rituxan
Started | 16
Completed | 9
Not Completed | 7
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1
Not completed — Patient Request | 1
Not completed — Investigator Request | 1

BASELINE CHARACTERISTICS:
Population: ITT population
Arm/Group | Gemzar + Novantrone + Rituxan
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 16
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (CR + PR)
Description: Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD.
Time Frame: 2 years
Population: Evaluable Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemzar + Novantrone + Rituxan
Number analyzed (Participants) | 15
percentage of participants | 46.7 [21.3 to 73.4]

2. Secondary Outcome: Duration of Response
Description: The duration of response is measured from the time measurement criteria are first met for CR/PR until the first date that recurrent or progressive disease is objectively documented.
  CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD.
Time Frame: From date of randomization until the date of first documented progression or the date of death from any cause, whichever came first, assessed up to 33 months.
Population: For patients who achieve a major objective response (CR or PR) the time to response will be assessed as the date of registration to the date of response.
Measure: Median (Full Range); unit: months
Arm/Group | Gemzar + Novantrone + Rituxan
Number analyzed (Participants) | 7
months | 7.9 [4.8 to 31.3]

3. Secondary Outcome: Overall Survival (OS) Rate at 1 Year
Description: OS is measured from the date of randomization to the date of death for a dead patient. If a patient is still alive or is lost to follow up, the patient will be censored at the last contact date.
Time Frame: 1 year.
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Probability of Survival
Arm/Group | Gemzar + Novantrone + Rituxan
Number analyzed (Participants) | 16
Probability of Survival | 0.57 [0.28 to 0.78]

4. Secondary Outcome: Progression-free Survival Rate at 1 Year.
Description: PFS is measured from the date of randomization to the date of first documented disease progression or date of death, whichever comes first. If a patient neither progresses nor dies, this patient will be censored at last contact date.
Time Frame: 1 year.
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Probability of Progression-free Survival
Arm/Group | Gemzar + Novantrone + Rituxan
Number analyzed (Participants) | 16
Probability of Progression-free Survival | 0.54 [0.24 to 0.77]

ADVERSE EVENTS:
Time Frame: During the whole treatment period, up to 30 days following last dose.
Description: For treated patients only, assessed at each treatment visit.
Arm/Group | Gemzar + Novantrone + Rituxan
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemzar + Novantrone + Rituxan (N=15)
CACHEXIA (General disorders) | 1 (1)
FEVER (General disorders) | 2 (3)
PAIN ABDO (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemzar + Novantrone + Rituxan (N=15)
ABDO ENLARGE (Gastrointestinal disorders) | 1 (1)
ALLERG REACT (Immune system disorders) | 2 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 (3)
ANEMIA (Blood and lymphatic system disorders) | 13 (49)
ANOREXIA (Gastrointestinal disorders) | 7 (10)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
ASTHENIA (General disorders) | 14 (35)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BILIRUBINEM (Metabolism and nutrition disorders) | 1 (1)
BUN INC (Metabolism and nutrition disorders) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
CHILLS (General disorders) | 2 (4)
CONSTIP (Gastrointestinal disorders) | 6 (7)
COUGH INC (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CREATININE INC (Metabolism and nutrition disorders) | 1 (1)
DEHYDRAT (Gastrointestinal disorders) | 1 (1)
DEPRESSION (General disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 2 (3)
DIZZINESS (Nervous system disorders) | 3 (3)
DRY MOUTH (Gastrointestinal disorders) | 3 (3)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 3 (5)
EDEMA PERIPH (Blood and lymphatic system disorders) | 1 (4)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
FEVER (General disorders) | 3 (3)
FLATUL (Gastrointestinal disorders) | 1 (1)
FLU SYND (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HEADACHE (General disorders) | 1 (2)
HEMATURIA (Renal and urinary disorders) | 1 (1)
HYPERGLYCEM (Metabolism and nutrition disorders) | 2 (4)
HYPERURICEM (Metabolism and nutrition disorders) | 1 (1)
HYPOCALCEM (Metabolism and nutrition disorders) | 2 (3)
HYPONATREM (Metabolism and nutrition disorders) | 1 (1)
HYPOPROTEINEM (Metabolism and nutrition disorders) | 2 (4)
HYPOVOLEM (Metabolism and nutrition disorders) | 1 (1)
INFECT (Infections and infestations) | 2 (2)
INSOMNIA (General disorders) | 1 (1)
LAB TEST ABNORM (Metabolism and nutrition disorders) | 1 (2)
LDH INC (Metabolism and nutrition disorders) | 2 (2)
LEUKOPENIA (Blood and lymphatic system disorders) | 9 (50)
MUCOUS MEM DIS (Skin and subcutaneous tissue disorders) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 9 (15)
NEUTROPENIA (Blood and lymphatic system disorders) | 15 (64)
PAIN (General disorders) | 3 (3)
PAIN ABDO (Gastrointestinal disorders) | 2 (2)
PAIN BONE (Musculoskeletal and connective tissue disorders) | 1 (3)
PAIN CHEST SUBSTERN (Investigations) | 1 (1)
PALLOR (Investigations) | 1 (2)
PHOSPHATASE ALK INC (Metabolism and nutrition disorders) | 1 (1)
PLAT ABNORM (Investigations) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 3 (4)
RECTAL DIS (Gastrointestinal disorders) | 1 (1)
RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
STOMATITIS (Respiratory, thoracic and mediastinal disorders) | 1 (2)
SWEAT (General disorders) | 2 (4)
TASTE PERVERS (Gastrointestinal disorders) | 3 (3)
THROMBOCYTHEM (Blood and lymphatic system disorders) | 1 (3)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 12 (63)
VASODILAT (Investigations) | 1 (1)
VOMIT (Gastrointestinal disorders) | 2 (3)
WEIGHT DEC (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No